CLINICAL TRIAL: NCT03648554
Title: A Multicentre Controlled and Randomized Study Assessing the Effect of Dulaglutide add-on to Dietary Reinforcement Versus Dietary Reinforcement Alone in Patients With Type 2 Diabetes and Carriers of a Non-alcoholic Steatohepatitis
Brief Title: Researching an Effect of GLP-1 Agonist on Liver STeatosis (REALIST)
Acronym: REALIST
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-002162-38; PSS2018/REALIST-GUERCI/AS (Other: sponsor code)
Record Dates: First submitted 2018-07-27; First posted 2018-08-27 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Type 2; NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease | interventions — dulaglutide

STUDY DESIGN:
Intervention Model Description: open, prospective, randomized, controlled study
Who Masked: Outcomes Assessor
Masking Description: Only centralized reading by the pathologist of the hepatic histology of the liver puncture biopsy (LPB) will be carried out in blinded procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dulaglutide (TRULICITY®) 1.5 mg (Experimental): dulaglutide (TRULICITY®) subcutaneous administration, one weekly injection, in a dose of 1.5 mg of dulaglutide for 52 weeks in combinaison with reinforced dietary monitoring as same as control group.
  Interventions: Drug: dulaglutide (TRULICITY®) 1.5 mg; Other: reinforced dietary monitoring
- reinforced dietary monitoring (Sham Comparator): reinforced dietary monitoring with frequent dietary consultations, based on American Heart Association (AHA) recommendations
  Interventions: Other: reinforced dietary monitoring

INTERVENTIONS:
Drug: dulaglutide (TRULICITY®) 1.5 mg — dulaglutide (TRULICITY®) 1.5 mg subcutaneous administration, one weekly injection over 52 weeks of treatment
  Arms: dulaglutide (TRULICITY®) 1.5 mg
Other: reinforced dietary monitoring — moderate caloric restriction individually adjusted according to the ideal weight and activity level, encouraging regular physical activity (about 30 minutes per day or 150-200 min per week)

SUMMARY:
GLP-1 analogues represent new treatments in diabetes that cause weight loss. Their effect on NASH in humans is unknown. A decrease in Alanine Aminotransferase (ALT) has been reported in pooled Exenatide/Placebo and Liraglutide/Placebo studies. More recently, LEAN study has shown that Liraglutide will result in improvements in liver histology in patients with NASH. It should be of high interest to investigate the effect of another GLP-1 Agonist as effective as Liraglutide, i.e. Dulaglutide in NASH.

Dulaglutide is one of the five GLP-1 receptor agonists approved for type 2 diabetes mellitus (T2DM). It is an effective treatment because it is dosed once-weekly, provides HbA1c reduction similar to Liraglutide, weight reduction similar to Exenatide, and has an adverse effect profile similar to other GLP-1 receptor agonists. Reduction in body weight was observed in patients treated with Dulaglutide, irrespective of nausea and/or vomiting.The search for a direct effect of Dulaglutide on liver fat overload in patients with type2 diabetes is required before considering the effectiveness of this treatment in NASH in diabetic populations. No current GLP-1 study has been designed with a control group with the same weight loss than as in the treatment group.

Primary objective: The investigators aim to study the effect of Dulaglutide 1.5 mg (TRULICITY®) add-on to dietary reinforcement after 52 weeks of treatment, on the improvement of liver histology compared to dietary reinforcement alone in patients with type 2 diabetes and carriers of non-alcoholic steatohepatitis.

Secondary objectives:

* After 52 weeks of treatment, to assess the effect of dulaglutide (TRULICITY®) add-on to dietary reinforcement on Fibrosis score, Transaminase levels, body composition as measured by dual energy X-ray absorptiometry, lipid profile, glycemic control and weight. The effect of the treatment will also be assessed on quality of life.
* At 24 weeks after completion of the treatment, to assess the sustainability of dulaglutide (TRULICITY®) treatment add-on to dietary reinforcement on ALT and AST rates as well as on weight.

DETAILED DESCRIPTION:
This is a multicentre, open, prospective, randomized, controlled dietary reinforcement study.

* Treatment Group: dulaglutide (TRULICITY®) subcutaneous administration, one weekly injection, in a dose of 1.5 mg of dulaglutide in combinaison with reinforced dietary monitoring as same as control group.
* Control group: reinforced dietary monitoring with frequent dietary consultations, based on AHA recommendations:

All patients are monitored in the same way for dietary reinforcement.

The study will be conducted over the course of 80 weeks in 3 periods (13 visits):

* Period I: Run-in phase of 4 weeks
* Period II: Treatment phase of 52 weeks
* Period III: Follow-up phase of 24 weeks. The patient must return to the study centre to assess whether the response to treatment is time-dependent.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, < 75 years
* Patients with moderately controlled type 2 diabetes under oral antidiabetic drugs (OADs) (i.e. biguanides, sulfonylureas, glinides, alpha-glucosidase inhibitors) at a stable dose since at least 3 months. Standard basal insulin treatments for at least 6 months before inclusion are allowed in addition to predefined authorized OADs.
* 7.0%≤HbA1c≤ 9.0% confirmed in two assays over the last six months
* 25 <BMI <40 kg/m2
* Patients carriers of confirmed stable non-alcoholic steatohepatitis diagnosed by liver biopsy dating less than six months, with a NAS score ≥ 4 with at least 1 point in each of the categories (steatosis, ballooning and lobular inflammation) and with a fibrosis score greater than stage 1 fibrosis but less than stage 4 fibrosis
* Stable weight during the six months prior to inclusion, i.e. the change in weight must not exceed 5% in the last six months since the last liver puncture biopsy (LPB).
* Person volunteered to participate in the study, informed about study organization and having signed the consent form
* Person affiliated to or beneficiary of a social security plan
* Person undergone the medical examination adapted to research

  * At randomization: The diagnosis and the stage of non-alcoholic steatohepatitis must be confirmed after centralized reading of the hepatic histology of the liver puncture biopsy (LPB) performed within six months prior to inclusion, by a pathologist designated for the study.

Exclusion Criteria:

* Patients who received a treatment with a GLP-1 agonist, SGLT2 inhibitors, Thiazolidinediones (TZDs), hepatoprotective drugs such as silymarine (Legalon®) or Ursodeoxycholic acid (Cholurso®, Delursan®, Ursolvan®), vitamin E or Betaine during the six months prior to inclusion (3 months before the reference biopsy). Any treatment with DPP-4 inhibitors should be stopped on inclusion.
* Patients receiving rapid or short-acting mealtime insulin or premixed insulin in the last 6 months before screening visit
* Type 1 Diabetes
* Patients with idiopathic hemochromatosis
* Patients carriers of hepatitis B or C
* Terminal renal impairment (calculated clearance < 15 ml/min according to the CKD-EPI formula)
* Class III or IV congestive heart failure according to the NYHA classification
* Chronic alcoholism. The investigator while interviewing the patient at the baseline visit assesses alcohol consumption. This consumption must be limited to 30g/day of alcohol for men and 20g/day of alcohol for women
* Hepatic fibrosis with a Kleiner score ≥ F3 (for a score = F3, patients with a platelet count > 120,000 and an albumin concentration > 35 g/l can be included)
* Patients with gastrointestinal bleeding
* History of acute or chronic pancreatitis
* Personal or family history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC), or personal history of non-familial medullary thyroid carcinoma
* Patients who had bariatric surgery
* Patients who received drug treatment for obesity, notably Orlistat, during the last 6 months
* Patients with eating disorders (anorexia nervosa, bulimia nervosa, binge-eating disorder) which may compromise the achievement of dietary reinforcement goals
* Patients with a known allergy or hypersensitivity to the study product or one of its excipients
* Any other condition deemed incompatible with the proper conduct of the study as determined by the investigator
* Patient having participated in another biomedical research with the taking of an experimental drug within 3 months prior to the screening visit or subject under an exclusion period for other biomedical research.
* Woman of childbearing age without effective contraception
* Person referred in articles L.1121-5, L.1121-7 and L.1121-8 of the Public Health Code:

  * Pregnant, parturient or breastfeeding woman
  * Minor person (non-emancipated)
  * Adult person under legal protection (any form of public guardianship)
  * Adult person incapable of giving consent
* Person deprived of liberty for judicial or administrative decision, Person under psychiatric care according to articles L. 3212-1 and L. 3213-1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Responder's proportion difference between the two groups (dulaglutide (TRULICITY®) on top of dietary reinforcement vs. dietary reinforcement alone) | after 52 weeks of treatment
  A responder is defined as having a histological improvement defined as the regression of non-alcoholic steatohepatitis (decrease of at least two points in the NASH Activity Score [NAS] measured on three components: steatosis, lobular inflammatory foci and hepatocyte ballooning) without worsening of fibrosis (defined by the stage of the Kleiner fibrosis classification) on liver histology obtained by liver puncture biopsy Score > 4 = NASH confirmed Score 3-4 = borderline Score < 3 = absence of NASH

SECONDARY OUTCOMES:
Fibrosis Kleiner score | after 52 weeks of treatment
  Mean Changes in Kleiner score of fibrosis with distribution of patients into 3 groups according to the evolution of the score: improvement, stability or worsening.
Fibrosis using Fibrotest score | after 52 weeks of treatment
  Mean changes in Fibrotest measurement (six markers dosage: ALT, total bilirubin, GGT, Apolipoprotein A1, alpha2-macroglobulin, haptoglobin)
Fibrosis marker parameter | after 52 weeks of treatment
  Hyaluronic acid serum rate
Changes in serum levels of liver enzymes ALT and AST | after 52 weeks of treatment
  ALT and AST levels
Changes in Lipid parameters | after 52 weeks of treatment
  * LDL-cholesterol value
  * HDL-cholesterol value
  * Triglycerides value
Improvement in the glycemic control | after 52 weeks of treatment
  Fasting glucose
overall glycemic control improvement | after 52 weeks of treatment
  HbA1c
Change in body composition assessed by dual-energy x-ray absorptiometry scans | after 52 weeks of treatment
  changes in fat mass
Change in quality of life | after 52 weeks of treatment
  Quality of Life, Obesity and Diet Scale (QOLOD rating scale questionnaire).Items were grouped in 5 dimensions: physical impact, psycho-social impact, sexual impact, comfort with food, diet experience. Each item of the QOLOD questionnaire was graded from 1 to 5 (1: always/enormously; 2: often/a lot; 3: sometimes/moderately; 4: rarely/a little; 5: never/not at all). score was then calculated for each dimension by adding together its constituent items. Scores obtained by adding up answers graded from 1 to 5 of all items per dimension were transformed to convert the lowest and highest score possible to 0 and 100 respectively. Hence the higher the score, the better the quality of life.
Change in weight | after 52 weeks of treatment
  variation in weight between the beginning and the end of treatment
ALT and AST levels | At 24 weeks after completion of the treatment
  The sustainability of dulaglutide (TRULICITY®) treatment on ALT and AST rates
Weight | At 24 weeks after completion of the treatment
  The sustainability of dulaglutide (TRULICITY®) treatment on weight

CONTACTS AND LOCATIONS:
Overall Officials: Bruno GUERCI, Principal Investigator — CHRU de Nancy
Locations (9):
- France (9):
  - CHU de CAEN, Caen
  - CHU de DIJON, Dijon
  - Chu Marseille, Marseille
  - CHRU de MONTPELLIER, Montpellier
  - CHU de REIMS, Reims
  - CHU de ROUEN, Rouen
  - CHU de TOULOUSE, Toulouse
  - CHRU de NANCY, Vandœuvre-lès-Nancy
  - G.H.M les Portes du Sud, Vénissieux

IPD SHARING:
Plan to Share IPD: No